CLINICAL TRIAL: NCT05125796
Title: Comparison of iv Paracetamol, iv Dexketoprofen and Topical Lidocaine in Scorpion Sting: a Placebo Randomized Controlled Trial
Brief Title: Analgesic Use for Pain Relief in Scorpion Sting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Adiyaman University Medical Faculty of Research and Training Hospital, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-5-1
Record Dates: First submitted 2021-11-02; First posted 2021-11-18 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Scorpion Stings
MeSH Terms: conditions — Scorpion Stings | interventions — Acetaminophen; dexketoprofen trometamol; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- paracetamol (Active Comparator): 1000 mg intravenous paracetamol
  Interventions: Drug: paracetamol
- Dexketoprofen Trometamol (Experimental): 50 mg intravenous Dexketoprofen Trometamol
  Interventions: Drug: Dexketoprofen Trometamol
- topical lidocaine (Experimental): %5 lidocaine 5 gr topical
  Interventions: Drug: Lidocaine topical
- placebo (Placebo Comparator): 100 mL intravenous normal saline+ placebo topical pomade
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paracetamol — 1000 mg intravenous paracetamol in 100 mL normal saline
  Other Names: Paracerol (paracetamol)
  Arms: paracetamol
Drug: Dexketoprofen Trometamol — 50 mg intravenous dexketoprofen Trometamol in 100 mL normal saline
  Other Names: Revafen(Dexketoprofen Trometamol)
  Arms: Dexketoprofen Trometamol
Drug: Lidocaine topical — Application of 5 gr of 5% topical lidocaine
  Other Names: Anestol pomade(lidocaine)
  Arms: topical lidocaine
Drug: Placebo — 100 mL intravenous normal saline infusion+ placebo topical pomade application
  Other Names: Placebo(intravenous normal saline+placebo topical pomade)
  Arms: placebo

SUMMARY:
In scorpion stings, patients mostly apply with the complaint of pain. Emergency physicians need to relieve this pain quickly.

DETAILED DESCRIPTION:
Aim: In this study, the analgesic efficacy of intravenous (IV) paracetamol, IV dexketoprofen trometamol and topical lidocaine will be compared in patients presenting with pain after scorpion sting.

Methods: This study is a double-blind, randomized, placebo-controlled study conducted in a tertiary emergency department. Adult patients who applied to the study with no systemic findings after scorpion sting and especially with pain will be randomly assigned to one of 4 groups: IV paracetamol, IV dexketoprofen trometamol, topical lidocaine or placebo. In order to determine the intensity of pain, Visual Analog Pain Score (VAS) will be measured at the time of admission to the emergency department, at the 30th minute and at the 60th minute. Afterwards, the VAS score changes between the groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Scorpion sting with pain
* The diagnostic criteria of Grade 1 for Scorpion sting

Exclusion Criteria:

* Patients who denied to give informed consent
* Taking analgesic treatment (ice application or drugs etc.) in the last 6 hours
* Any symptoms and findings of systemic toxicity of scorpion sting
* Pregnant women
* Hemodynamically unstable patients
* Known allergy to drugs of the study
* Patients with renal disease
* The cases that passed more than 6 hours after the bite

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change of the intensity of pain | 30 minutes and 60 minutes after the study drug administered
  Pain intense will be measured by 100 mm visual analog scale (Zero; no pain and 100 mm; the worst pain) after 30th and 60th minutes later after the study drug administered

SECONDARY OUTCOMES:
Adverse events | 60 minutes after the study drug administered
  60 minutes after the study drug administered
need to rescue medication | 60 minutes after the study drug administered
  60 minutes after the study drug administered

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gülaçtı, Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)